CLINICAL TRIAL: NCT05497986
Title: Conventional Low Flow Oxygenation Versus High Flow Nasal Cannula in Hypercapnic Respiratory Failure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hôpital de Verdun (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Verdun2022_01
Record Dates: First submitted 2022-08-08; First posted 2022-08-11 (Actual); Last update posted 2022-08-11 (Actual); Status verified 2022-08

CONDITIONS: Hypercapnic Respiratory Failure; Acute Copd Exacerbation
Keywords: High Flow Nasal Cannula; High Flow Nasal Insufflation; High Flow Oxygen Therapy; High Flow Oxygenation
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Due to the nature of the intervention, nor the participants, nor the treating physicians, nor the investigator can be blinded. However, the outcomes will be analyzed an independent statistician blinded to the treatment assignments.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Flow Nasal Cannula (Experimental)
  Interventions: Device: High flow nasal cannula
- Conventional Oxygenation with low flow cannula (Active Comparator)
  Interventions: Device: Conventional low flow oxygenation

INTERVENTIONS:
Device: High flow nasal cannula — HFNC with the maximum tolerated flow (up to 60 L/min). Titration of supplemental oxygen to a SpO2 between 88 - 92%.
  Other Names: High flow oxygenation; High flow oxygen therapy
  Arms: High Flow Nasal Cannula
Device: Conventional low flow oxygenation — Conventional oxygenation through nasal prongs or a facemask, with supplemental oxygen titrated to a SpO2 between 88 - 92%.
  Arms: Conventional Oxygenation with low flow cannula

SUMMARY:
Current evidence suggests a mechanistic and physiological rationale for the use of high flow nasal cannula (HFNC) in acute respiratory hypoxemic failure (AHRF) based on physiological studies in airway models, healthy volunteers and patients with Chronic Obstructive Respiratory Disease (COPD). This is supported by observational studies in patients with AHRF with reductions in a range of respiratory and other physiological parameters. Observational studies also suggest similar intubation rates and lower failure rates with HFNC when compared to non-invasive ventilation (NIV) with improved patient acceptance and tolerance for HFNC.

The role of HFNC is less clear in acute hypercapnic respiratory failure. Although non-invasive ventilation is the recommended treatment, it is associated with discomfort, and a significant proportion (up to 25% in some reports) cannot tolerate non-invasive ventilation. Observational reports and limited data from randomized controlled trials suggests that HFNC is effective in treating patients with hypercapnic respiratory failure.

We designed this trial to assess whether early application of HFNC in patients with non-severe hypercapnic respiratory failure can correct barometric abnormalities, and prevent progression to non-invasive ventilation or tracheal intubation and mechanical ventilation.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients > 18 years of age
* Acute Hypercapnic respiratory failure with pH < 7.35 and pCO2 > 45 mmHg

Exclusion Criteria:

* Pregnant or Breast-Feeding
* Patients who cannot read and understand French or English
* Hypercapnia secondary to a drug toxicity or non-pulmonary aetiology
* Hypercapnia secondary to exacerbation of asthma
* Contraindication to NIV
* Contraindication to HFNC
* Not for escalation to NIV based on a ceiling of care
* pH < 7.15
* GCS 8 or less
* Shock defined as systolic < 90 mmHg or a reduction by 20mmHg from usual systolic BP despite volume resuscitation
* Respiratory or cardio-respiratory arrest
* Any other indication that requires immediate invasive/non-invasive mechanical ventilation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2022-10 (Estimated); Primary Completion 2024-01 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients progressing to NIV in each cohort | 6 hours

SECONDARY OUTCOMES:
Venous blood gas PCO2 | 1 hour, 6 hours, and 24 hours
Venous blood gas pH | 1 hour, 6 hours, and 24 hours
Respiratory rate | 1 hour, 6 hours, 24 hours, and daily until study completion
  Number of breaths per minute, as documented in the medical chart
Heart rate | 1 hour, 6 hours, 24 hours, and daily until study completion
  Number of heart beats per minute, as documented in the medical chart
Mean arterial pressure | 1 hour, 6 hours, 24 hours, and daily until study completion
  Mean arterial pressure, as documented in the medical chart
Incidence of intubation | Up to 90 days after enrolment, or until hospital discharge
Admission to the intensive care unit | Up to 90 days after enrolment, or until hospital discharge
In-hospital mortality | Up to 90 days after enrolment, or until hospital discharge
Intensive care unit length of stay | Up to 90 days after enrolment, or until discharge from the intensive care unit
Hospital length of stay | Up to 90 days after enrolment, or until hospital discharge
Patient comfort | 1 hour, 6 hours, 24 hours, and daily until cessation of oxygen therapy, up to a maximum of 7 days
  Level of comfort assessed on a visual analogue scale by the patient
Shortness of breath | 1 hour, 6 hours, 24 hours, and daily until cessation of oxygen therapy, up to a maximum of 7 days
  Severity of the shortness of breath assessed on a visual analogue scale by the patient

CONTACTS AND LOCATIONS:
Overall Officials: Ivan Pavlov, M.D., Principal Investigator — CIUSSS-Centre-Sud-de-l'Île-de-Montréal
Locations (3):
- Canada (3):
  - CISSS-de-la-Montérégie-Centre, Longueuil, Quebec
  - CIUSSS de l'Est-de-l'ïle-de-Montréal, Montreal, Quebec
  - Hôpital de Verdun, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: Yes
Data may be shared to researchers who will request it, based on reasonable research objectives, ethical approval if needed, and signing of a data sharing agreement by the relevant institutions.